CLINICAL TRIAL: NCT02405130
Title: Impact of intRacoronary adrEnaline on Myocardial reperfuSion in STEMI paTients With Persistent Impaired cORonary Flow After pErcutaneous Coronary Intervention: the RESTORE-SIRIO Randomized Controlled Trial
Brief Title: The RESTORE-SIRIO Randomized Controlled Trial
Acronym: RESTORE-SIRIO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: SIRIO MEDICINE (Unknown)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Klinik für Kardiologie, Pneumologie und Angiologie, Heinrich-Heine University, Duesseldorf
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RESTORE-SIRIO
Record Dates: First submitted 2015-03-24; First posted 2015-04-01 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Percutaneous Coronary Intervention; No-reflow Phenomen; Acute ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- epinephrine (Active Comparator): intracoronary epinephrine is two ampoules each of 1:1000 epinephrine (1 μg/mL) diluted into 100 mL of normal saline (to 20 μg/mL epinephrine solution); a 5 ml syringe prepared will then contain 100 μg
  Interventions: Other: intracoronary epinephrine
- no intracoronary epinephrine (Other): no epinephrine
  Interventions: Other: no intracoronary epinephrine

INTERVENTIONS:
Other: intracoronary epinephrine — after failure of standard therapy patients will treated with epinephrine
  Arms: epinephrine
Other: no intracoronary epinephrine — patients will receive standard therapy only
  Arms: no intracoronary epinephrine

SUMMARY:
Primary percutaneous coronary intervention (PPCI) is the preferred reperfusion strategy for treating acute ST-segment elevation myocardial infarction (STEMI). The main goals are to restore epicardial infarct-related artery patency and to achieve microvascular reperfusion as early as possible. No-reflow is the term used to describe inadequate myocardial perfusion of a given coronary segment without angiographic evidence of persistent mechanical obstruction of epicardial vessels and it refers to the high resistance of microvascular blood flow encountered during opening of the infarct-related coronary artery.

Despite optimal evidence-based PPCI, myocardial no-reflow can still occur, negating many of the benefits of restoring culprit vessel patency, and is associated with a worse in-hospital and long-term prognosis. Several strategies have been tested to revert the no-reflow including the use of thrombectomy, glycoprotein IIb/IIIa inhibitors and the use of intracoronary adenosine, but none has been demonstrated to effectively counteract the phenomenon.

The trial aims to show the effect of the administration of intracoronary adrenalin on myocardial reperfusion assessed by magnetic resonance in patients with STEMI undergoing PCI and with persistent coronary angiographic The Thrombolysis in Myocardial Infarction (TIMI) 0-1 flow during the interventional procedure after failure of standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* presentation within 6-7 h of symptom onset of STEMI
* eligibility for reperfusion by primary-PCI
* TIMI flow grade 0-1 during the interventional procedure in the culprit vessel after the initial opening of the vessel with the coronary wire

Exclusion Criteria:

* evident clinical arrhythmias (ventricular tachycardia/ventricular fibrillation)
* evidence of coronary dissection or spasm
* Parkinson symptoms
* closed angle glaucoma
* thyroid disorders
* known history to hypersensitivity to the drug
* pregnancy
* stage 4 or 5 CKD (eGFR <30 mL/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
myocardial infarct size (% total LV mass) | 48-72 hours post intervention
  cMRI parameters: myocardial infarct size (% total LV mass)

SECONDARY OUTCOMES:
Incidence and extent of microvascular obstruction | 48-72 hours and 30 days post intervention
  cMRI parameter
Myocardial salvage index (MSI) | 48-72 hours and 30 days post intervention
  cMRI parameter
Intra-myocardial haemorrhage (IMH) | 48-72 hours and 30 days post intervention
  cMRI parameter
LV ejection fraction (LVEF) and volumes | 48-72 hours and 30 days post intervention
  cMRI parameter
Thrombolysis in Myocardial Infarction (TIMI) flow grade) | 48-72 hours post intervention
  Angiographic markers
Myocardial blush grade (MBG) | 48-72 hours post intervention
  Angiographic markers
Computer-assisted myocardial blush quantification using the software 'Quantitative Blush Evaluator' (QuBE) | 48-72 hours post intervention
  Angiographic markers
Degree of ST segment resolution on ECG | 48-72 hours post intervention

OTHER OUTCOMES:
creatine kinase and troponin I release | 48-72 hours post intervention
major cardiovascular events (MACE) | 30 days post intervention
  death, need for Target Lesion Revascularization, recurrent myocardial infarction (MI), new or worsening heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Eliano P Navarese, MD, PhD, FESC, Study Director — Division of Cardiology, Pulmonary Disease and Vascular Medicine, Heinrich-Heine University Dusseldorf
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

REFERENCES:
- See also: Related Info — http://www.uniklinik-duesseldorf.de/kardiologie
- See also: Related Info — http://siriomedicine.com/